CLINICAL TRIAL: NCT04481828
Title: Comparison With Open and Totally Laparoscopic Gastrectomy for Gastric Cancer in a Low Volume Center
Brief Title: Comparison With Open and Totally Laparoscopic Gastrectomy for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Yuksel, M.D. Department of Gastroenterological surgery,Principal Investigator, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2019-98
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- open gastrectomy: The first group (Group 1; n: 30) consisted of patients who underwent open surgery
  Interventions: Procedure: gastrectomy
- laparoscopic gastrectomy: The second group (group 2; n:30) consisted of patients who underwent laparoscopic gastrectomy
  Interventions: Procedure: gastrectomy

INTERVENTIONS:
Procedure: gastrectomy — gastric resection with lymph node dissection(D1+,D2) for stomach cancer.

SUMMARY:
In gastric cancer, laparoscopic gastrectomy is commonly performed in Asian countries. In other regions where tumor incidence is relatively low and patient characteristics are different, developments in this issue have been limited. In this study, the investigators aimed to compare the early results for patients who underwent open or laparoscopic gastrectomy for gastric cancer in a center in Turkey.

DETAILED DESCRIPTION:
The patients who were operated in Kocaeli Derince Training and Research Hospital between January 2014 and January 2019 consecutively due to gastric cancer were analyzed. The diagnosis was made by upper gastrointestinal endoscopy and endoscopic biopsy. Clinical staging was done using contrast computed tomography (CT). Positron emission tomography (PET) was used in patients with suspected metastasis.The patients were divided into two groups according to the technique applied (open, laparotomy). The first group (Group 1; n: 30) consisted of patients who underwent open surgery, and the second group (Group 2, n: 30) laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer(adenocarcinoma) proven biopsy
* Operated by same surgical team
* Presence of distant metastasis

Exclusion Criteria:

* Patients who underwent palliative resection
* operated by a different surgical team
* ASA score: 4

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were operated in Kocaeli Derince Training and Research Hospital between January 2014 and January 2019 consecutively due to gastric cancer.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Age | 2014-2019
  year
Body mass index | 2014- 2019
  kg/m2
Previous abdominal surgery status | 2014-2019
  yes or no
Comorbidity status | 2014 -2019
  present or absent
Neoadjuvant therapy status | 2014-2019
  present or absent
American Society of Anesthesiologists (ASA) score | 2014-2019
  1,2,3,4
Gender | 2014-2019
  male or female
Surgical technique | 2014-2019
  open or laparoscopic
Tumor localization | 2014 - 2019
  proximal, middle, lower
Gastrectomy type | 2014 - 2019
  total, subtotal
Lymph node dissection type | 2014 - 2019
  D1+, D2
Operation time | 2014 - 2019
  minute
Blood loss | 2014 - 2019
  ml
Complication (Clavien-Dindo Classification) | 2014 - 2019
  1,2,3 A,3 B,4 A,4 B,5 (according to Clavien-Dindo Classification)
30-day mortality | 2014 - 2019
  present or absent
Number of harvested lymph node | 2014 - 2019
  number
Resection margin status | 2014 - 2019
  positive or negative
Tumor stage (American Joint Committee on Cancer 8th Edition) | 2014 - 2019
  0,1,2 A,2 B,3,4 A, 4 B (According to American Joint Committee on Cancer 8th Edition)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Derince Training and research Hospital, Kocasinan, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okabe H, Tsunoda S, Obama K, Tanaka E, Hisamori S, Shinohara H, Sakai Y. Feasibility of Laparoscopic Radical Gastrectomy for Gastric Cancer of Clinical Stage II or Higher: Early Outcomes in a Phase II Study (KUGC04). Ann Surg Oncol. 2016 Aug;23(Suppl 4):516-523. doi: 10.1245/s10434-016-5383-0. Epub 2016 Jul 11. PMID 27401443
- [Background] van der Wielen N, Straatman J, Cuesta MA, Daams F, van der Peet DL. Short-term outcomes in minimally invasive versus open gastrectomy: the differences between East and West. A systematic review of the literature. Gastric Cancer. 2018 Jan;21(1):19-30. doi: 10.1007/s10120-017-0747-0. Epub 2017 Jul 20. PMID 28730391
- [Background] Haverkamp L, Ruurda JP, Offerhaus GJ, Weijs TJ, van der Sluis PC, van Hillegersberg R. Laparoscopic gastrectomy in Western European patients with advanced gastric cancer. Eur J Surg Oncol. 2016 Jan;42(1):110-5. doi: 10.1016/j.ejso.2015.09.018. Epub 2015 Oct 22. PMID 26603678